CLINICAL TRIAL: NCT03388489
Title: The Physiological and Psychological Effect of Mind-Body Walking Exercise for Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Mind-Body Walking Exercise for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201312004RIND
Record Dates: First submitted 2017-12-08; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Exercise; Anxiety; Depression; Dyspnea; Quality of Life; Heart Rate Variability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Anxiety Disorders; Depression; Dyspnea

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Body Walking (Experimental): breathing, walking and meditation
  Interventions: Behavioral: Mind-Body Walking
- Usual care (No Intervention): maintain their daily activity

INTERVENTIONS:
Behavioral: Mind-Body Walking — walking, breathing, and mindfulness
  Arms: Mind-Body Walking

SUMMARY:
Mind-body exercise improves symptom of negative moods, dyspnea and quality of life in chronic diseases, but these improvements for chronic obstructive pulmonary disease (COPD) are unproven. This study aims to examine the effects of dyspnea, exercise capacity, heart rate variability(HRV), anxiety, depression, interoceptive awareness, quality of life(QoL) in patients with COPD across a three-month mind-body exercise program.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive disease characterized by airflow limitation, has a high prevalence of morbidity and mortality, and results in negative physical, psychological, and quality of life (QoL) impacts. Patients with COPD typically experience dyspnea, exercise intolerance, autonomic dysfunction, anxiety, depression, and poor QoL. Mind-body intervention with walking, breathing, and mindfulness is beneficial for the health of patients with COPD. However, the result of mind-body walking intervention for patients with COPD is not clear. Thus, this study will evaluate the effects of mind-body walking exercise (MBWE) on the physical psychological wellbeing and QoL of patients with COPD.

This study will be a randomized controlled trial. Data will collect from the pulmonary clinics of a medical center in northern Taiwan. The participants will recruit and randomly assign into the MBWE group or the control group. Participants in the control group will receive their usual care. Participants in the MBWE group will receive not only their usual care but also a MBWE program, consisting of walking, breathing, and mindfulness activities, for 30 min per day, 5 days per week, for 8 weeks. Data will collect at baseline and follow up on week 4 (WK 4), week 8 (WK 8), and week 12 (WK12). The primary outcome is dyspnea using modified Borg scale. The secondary outcomes are dyspnea in daily life using modified Medical Research Council (mMRC), exercise capacity using six minute walk distance (6MWD), Heart rate variability (HRV), anxiety and depression using the Hospital Anxiety and Depression scale (HADS), interoceptive awareness using the Multidimensional Assessment of Interoceptive Awareness- Chinese version (MAIA-C), QoL using COPD Assessment Tes (CAT). The independent t-test and Chi-square test were used to examine the homogeneity of the demographic characteristics of two groups. Generalized estimating equations were used to examine the data from repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

1.mild to severe COPD

Exclusion Criteria:

1. Patients visited the emergency room or were hospitalized previous month;
2. Long-term oxygen therapy;
3. Atrial fibrillation;
4. Severe cognitive impairment;
5. Great than class II heart failure as defined by the New York Heart Association functional classification in previous six months;
6. Pacemaker were excluded;
7. Received cancer treatment
8. Participated in other exercise trials

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2015-08-13 (Actual); Study Completion 2015-08-13 (Actual)

PRIMARY OUTCOMES:
Change of modified Borg scale for dyspnea level | Baseline and follow up on Week 4, 8, and 12.
  The modified Borg scale is a visual tool ranging from 0 (not noticeable) to 10 (maximum dyspnea).

SECONDARY OUTCOMES:
Heart rate variability (HRV) | Baseline and follow up on Week 4, 8, and 12.
  An HRV monitor (8Z11, Enjoy Research Inc., Taiwan) was used. Participants were instructed to avoid caffeine or other stimulants food before the measurement and to breathe normally in a seated position at rest during the five-minute measurement. Selected parameters of HRV were standard deviation of all NN intervals (SDNN), power in low frequency range (LF, 0.04-0.15 Hz), power in high frequency range (HF, 0.15-0.40 Hz) and LF/HF ratio (Camm et al., 1996). SDNN represented the autonomic function (141±39 for normal value); LF represented both vagal and sympathetic activity (1170±416 for normal value); HF represented vagal control (975±203 for normal value); and LF/HF ratio represented sympatho-vagal balance (0.5~2.5 for normal value) (Camm et al., 1996). The measurements of HRV were taken between 9 a.m. and 5 p.m. to minimize the effect of circadian rhythm on heart rate measurements. The raw data of the measures were used in the study.
Hospital anxiety and depression scale (HADS) for anxiety and depression | Baseline and follow up on Week 4, 8, and 12.
  Hospital anxiety and depression scale (HADS) consists seven items for anxiety and seven items for depression. Four scores (0-3) were designed for each item, with higher score indicating higher anxiety and depression. The score of anxiety or depression domain below 8 indicates no anxiety or depression.
The Chinese version multidimensional assessment of interoceptive awareness (MAIA-C) for interoceptive awareness | Baseline and follow up on Week 4, 8, and 12.
  The Chinese version multidimensional assessment of interoceptive awareness (MAIA-C) included five scales of emotional awareness, attention regulation, body listening, noticing, and self-regulation. Response was rated on six-point Likert scale from 0 (never) to 5 (always), higher scores represented greater interoceptive awareness.
Six-minute walk distance for exercise capacity | Baseline and follow up on Week 4, 8, and 12.
  Six-minute walk distance (6MWD) from the six-minute walk test (American Thoracic Society 2002) was tested. Participants were encouraged to walk as far as possible in six minutes along a flat straight corridor, but they could stop or slow down during the test, if necessary. Longer distances represent greater exercise capacity.
modified Medical Research Council (mMRC) for perception of dyspnea in daily life | Baseline and follow up on Week 4, 8, and 12.
  The modified Medical Research Council (mMRC has five score (0～4), with 0 of "I get breathless when strenuous exercise", and 4 of "I get breathless when dressing or leaving the house". A higher score means higher dyspnea.
COPD assessment test (CAT) for quality of life | Baseline and follow up on Week 4, 8, and 12.
  COPD assessment test (CAT) composes of eight items, including the levels of cough, phlegm (mucus), chest tight, walk up a hill or one flight of stair, limited of activities at home, confident of leaving home, sleep status, and energy. Each item scores 0~5, and a total score is 0~40. A higher score means worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Lien Lin, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin FL, Yeh ML, Lai YH, Lin KC, Yu CJ, Chang JS. Two-month breathing-based walking improves anxiety, depression, dyspnoea and quality of life in chronic obstructive pulmonary disease: A randomised controlled study. J Clin Nurs. 2019 Oct;28(19-20):3632-3640. doi: 10.1111/jocn.14960. Epub 2019 Jun 28. PMID 31192478